CLINICAL TRIAL: NCT04999878
Title: A Prospective Clinical Study of Ruxolitinib Phosphate Tablets and Etoposide Combined With DDGP Regimen (RUE-DDGP) in Induction Therapy of T/NK Cell Lymphoma-associated Hemophagocytic Syndrome.
Brief Title: A Prospective Clinical Study of Ruxolitinib and Etoposide Combined With DDGP Regimen (RUE-DDGP) in Induction Therapy of T/NK Cell Lymphoma-associated Hemophagocytic Syndrome.
Acronym: RUE-DDGP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx20210601
Record Dates: First submitted 2021-08-03; First posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Hemophagocytic Syndrome; T/NK-Cell Lymphoma
Keywords: ruxolitinib; Lymphoma-associated Hemophagocytic Syndrome; Etoposide; Dexamethasone; Pegaspargase; Gemcitabine; cis-platinum
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Lymphoma, Extranodal NK-T-Cell | interventions — ruxolitinib; Etoposide; Dexamethasone; Gemcitabine; pegaspargase; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): All enrolled patients will receive a regimen containing Ruxilitinib, Etoposide, Dexamethasone, Gemcitabine, Pasparase and Platinum for 28 days. The specific medication is as follows:
  Ruxilitinib 10 mg, bid, d1-28, P.O. Etoposide 100mg per week, two weeks, ivgtt Dexamethasone, 15mg/(m²·d)，d1-12，10 mg/ (m²·d) ，d13-14，5 mg/ (m²·d) ，d15-21，2.5mg/(m²·d)，d22-28，ivgtt or P.O.
  Gemcitabine, 0.5 g/m², d8, ivgtt Pegaspargase, 2500IU/m², d9, im Platinum, 20mg/m² d10 d11, ivgtt After the treatment, patients will be given disease specific chemotherapy regimen to treat lymphoma according to patient's different lymphoma subtype.
  Interventions: Drug: Ruxolitinib, Etoposide, Dexamethasone, Gemcitabine, Pegaspargase, cis-platinum

INTERVENTIONS:
Drug: Ruxolitinib, Etoposide, Dexamethasone, Gemcitabine, Pegaspargase, cis-platinum — All enrolled patients will receive a regimen containing Ruxilitinib, Etoposide, Dexamethasone, Gemcitabine, Pasparase and Platinum for 28 days. The specific medication is as follows:
  Ruxilitinib 10 mg, bid, d1-28, P.O. Etoposide 100mg per week, two weeks, ivgtt Dexamethasone, 15mg/(m²·d)，d1-12，10 mg/ (m²·d) ，d13-14，5 mg/ (m²·d) ，d15-21，2.5mg/(m²·d)，d22-28，ivgtt or P.O.
  Gemcitabine, 0.5 g/m², d8, ivgtt Pegaspargase, 2500IU/m², d9, im Platinum, 20mg/m² d10 d11, ivgtt After the treatment, patients will be given disease specific chemotherapy regimen to treat lymphoma according to patient's different lymphoma subtype.

SUMMARY:
To observe the efficacy and safety of Ruxolitinib and Etoposide combined with DDGP regimen ( cis-Platinum, Dexamethasone, Gemcitabine and Pegaspargase) in the first-line induction therapy of T cell lymphoma and NK/T cell lymphoma-associated hemophagocytic syndrome.

DETAILED DESCRIPTION:
This is an open, one-arm, prospective clinical collaborative study. This study is aimed to observe the efficacy and safety of the new combined therapy of Ruxolitinib and Etoposide combined with DDGP regimen ( cis-Platinum, Dexamethasone, Gemcitabine and Pegaspargase) in the first-line induction therapy patients with primary central nervous system lymphoma. A total of 30 patients plan to participate in the study. The primary endpoint is objective remission rate (ORR) of hemophagocytic syndrome, and the secondary endpoints include progression-free survival (PFS) , objective remission rate (ORR) of lymphoma, overall survival (OS), and adverse events(ADR).

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically proven T-cell lymphoma or NK/ T-cell lymphoma;
2. Comply with HLH-2004 diagnostic criteria;Hemophagocytic syndrome can be diagnosed when either of the following two criteria is met:

   A. Molecular diagnosis is consistent with hemophagocytic syndrome. Pathological mutations were found in known pathogenic genes related to hemophagocytic syndrome, such as PRF1, UNC13D, STX11, STXBP2, RAB27A, LYST, SH2D1A, BIRC4, ITK, AP3B1, MAGT1, CD27, etc.

   B. Meet 5 of the following 8 indicators I. Fever: The body temperature was > 38.5℃, lasting > for 7 days. II. Splenomegaly . III. Hemocytopenia (involving two or three lines of peripheral blood) : hemoglobin < 90g/L, platelet < 100×10^9/L, neutrophils < 1.0×10^9/L and not caused by reduced hematopoietic function of bone marrow.

   IV. Hypertriglyceridemia and/or hypofibrinogenemia: triglyceride > 3mmol/L or 3 standard deviations higher than the same age, fibrinogen < 1.5g/L or 3 standard deviations lower than the same age.

   V. Hemophagocytes are found in bone marrow, spleen, liver, or lymph nodes. VI.NK cell activity decreased or absent. VII. Elevated serum ferritin: ferritin ≥500μg/L. VIII. Elevated sCD25 (soluble interleukin-2 receptor).
3. Ages 14-75 years.
4. Expected survival of more than 1 week.
5. Patients with left ventricular ejection fraction > 50%, no major bleeding of active internal organs (digestive tract, lung, brain, etc.), and oxygenation index > 250.
6. Patients have good compliance with the planned treatment and follow-up, can understand the research process of this study and sign the written informed consent.

Exclusion Criteria:

1. Three or more drugs including ruxolitinb, etoposide, pemasparase, gemcitabine or cisplatin were used simultaneously in the previous 28 days.
2. Pregnant or lactating women and patients of reproductive age who refuse to take appropriate contraceptive measures during the course of this study. If the patient was male, they refused to use adequate contraception or sperm donation during the study period and for 3 months after the last study of lymphoma-related chemotherapy drugs.
3. Allergic to any medication in the program.
4. Grade III or IV heart disease based on the New York Heart Association (NYHA) score.
5. Major active bleeding of internal organs (including gastrointestinal bleeding, alveolar bleeding, intracranial bleeding, etc.).
6. Acute pancreatitis.
7. People infected with HIV (HIV antibody positive).
8. HBV DNA copy number is >10^4/ml in patients with acute or chronic active hepatitis B, and HBV DNA copy number is >10^4/ml in patients with acute or chronic active hepatitis C (HCV antibody positive, HCV RNA negative acceptable).
9. Participate in other clinical investigators.
10. The investigators identified patients who were not eligible for the study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR of hemophagocytic syndrome | 28 days
  Objective remission rate of hemophagocytic syndrome

SECONDARY OUTCOMES:
PFS | up to 24 months
  Progression-free survival
ORR of lymphoma | up to 24 months
  Objective remission rate of lymphoma
OS | up to 24 months
  Overall Survival
ADR | up to 24 months
  Adverse Reaction Rate

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chang, Pro.Dr., Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China